CLINICAL TRIAL: NCT01821417
Title: A Randomized Clinical Trial to Assess the Performance of MicroTextured Dental Implants With or Without a Machined Collar
Brief Title: Performance of MicroTextured Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Zimmer Dental (Industry)
Responsible Party: Principal Investigator, Michael Reddy, DMD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Z-11
Record Dates: First submitted 2013-03-13; First posted 2013-04-01 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2017-03-16 (Actual); Status verified 2017-01

CONDITIONS: Partially Edentulous Jaw
Keywords: dental implants; screw-vent dental implants
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microtextured dental implant (Experimental): Randomized for microtextured dental implant treatment
  Interventions: Device: Microtextured dental implant treatment
- Dental implant (Active Comparator): Randomized dental implant treatment with machined-collar implants
  Interventions: Device: Dental implant treatment

INTERVENTIONS:
Device: Microtextured dental implant treatment — Microtextured dental implant treatment will include a surgically inserted device implanted into edentulous areas of the jaw where natural teeth have been lost and adequate bone exists.
  Other Names: Screw-vent dental implant
  Arms: Microtextured dental implant
Device: Dental implant treatment — Treatment with dental implants; implants with a machined collar will be surgically implanted into edentulous areas of the jaw where natural teeth have been lost and adequate bone exists.
  Arms: Dental implant

SUMMARY:
The study will compare initial peri-implant bone healing and longitudinal osseointegration between a fully microtextured dental implant and an analogous implant with a smooth machined collar.

The investigators hypothesize the fully textured implant will result in less peri-implant crestal bone resorption than the implant with a machined collar.

DETAILED DESCRIPTION:
Zimmer dental has developed a microtextured tapered screw-vent implant design with a titanium skin that has been grit-blasted with hydroxyapatite particles resulting in an overall roughened surface, which, when compared to an implant with a machined (smooth) collar (narrow band around the top of the device) surface is thought to increase the apposition of osseous tissue integration and to promote epithelial attachment to the implant device.

ELIGIBILITY:
Inclusion Criteria:

1. Be a current registered University of Alabama at Birmingham (UAB)dental school patient
2. Existence of one or more missing teeth scheduled to be replaced with dental implants
3. Healthy enough to undergo proposed therapy without compromising existing health
4. Able to consent for their own inclusion
5. Able to read and understand the informed consent form
6. Demonstrated willingness to comply with protocol requirements and timeline

Exclusion Criteria:

1. Any health condition that in the opinion of the investigators may adversely affect bone healing
2. Any medication that in the opinion of the investigators may adversely affect bone healing
3. Any indication of an inability to make autonomous decisions
4. Reported pregnancy at the time of enrollment -

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-05; Primary Completion 2014-06 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas C. Geurs, DDS.MS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham School of Dentistry, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Microtextured Dental Implant | Dental Implant
Started | 37 | 31
Completed | 37 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Microtextured Dental Implant | Dental Implant | Total
Number analyzed (Participants) | 37 | 31 | 68
Age, Customized [Number; unit: participants]
  Greater than 19 years | 37 | 31 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 21 | 20 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 35 | 31 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 28 | 23 | 51
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 31 | 68

OUTCOME MEASURES:

1. Primary Outcome: Change in Millimeters of Bone Loss Surrounding the Implant Device
Description: Using radiographic images and image-processing software, measurements of bone height at the mesial and distal of each implant will be captured in millimeters.
Time Frame: Implant insertion, 12 months post-insertion
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Microtextured Dental Implant | Dental Implant
Number analyzed (Participants) | 37 | 31
millimeters | -0.35 (0.56) | -0.82 (0.70)

2. Secondary Outcome: Changes in Peri-implant Gingivitis Score
Description: Measurement of changes in peri-implant gingivitis score [Loe and Silness gingival index (GI)] after implant restoration
Time Frame: 1 year after placement
Population: No data was collected. Previously entered data was entered incorrectly.
Arm/Group | Microtextured Dental Implant | Dental Implant
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Millimeters of Periodontal Pocket Depth Surrounding the Dental Implant Device
Description: Probing pocket depth (PD) is measured from the mucosal sulcus to the depth of the pocket attachment after implant restoration.
Time Frame: 1 year after placement
Population: No data was collected. Previously entered data was entered incorrectly.
Arm/Group | Microtextured Dental Implant | Dental Implant
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Microtextured Dental Implant; Dental Implant: Serious adverse events are defined as life threatening events that occur during the course of the study treatment that may or may not be related to study protocols and procedures.
  Other adverse events are defined as non-life threatening events that are unexpected after the routine performance of the study protocols and procedures. These may or may not be related to the study protocols and procedures.
Arm/Group | Microtextured Dental Implant | Dental Implant
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/31
Other Adverse Events (participants affected / at risk) | 0/37 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes